CLINICAL TRIAL: NCT04136964
Title: Cross-cultural Adaptation and Validation of Arabic Version of the Core Outcome Measure Index (COMI) in Patients With Chronic Neck Pain
Brief Title: Cross-cultural Adaptation and Validation of Arabic Version of COMI in Patients With Chronic Neck Pain
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Aliaa Rehan Youssef, Assistant professor of Orthopedic Physical Therapy, Cairo University
Other Study IDs: SYahya
Record Dates: First submitted 2019-10-21; First posted 2019-10-23 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Chronic Neck Pain
Keywords: Neck pain; COMI; Quality of life; Questionnaire; Validity; Reliability; Patient-reported outcome measures
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients group: Patients who have pain located in the anatomical region of the neck for more than three months due to mechanical causes; with or without radiation to the head, trunk, and upper limbs. Posteriorly, pain may be present in the neck region from the superior nuchal line to the spine of the scapula and the side region down to the superior border of the clavicle and the suprasternal notch.
  Interventions: Other: Neck COMI

INTERVENTIONS:
Other: Neck COMI — Patients will be asked to fill a questionnaire booklet consisting of five patient-reported outcome measures twice within 14 days.
  Other Names: VAS, NDI, EQ-VAS, EQ-5D

SUMMARY:
PURPOSE:

To translate, validate and examine the psychometric properties of the Arabic version of the COMI in Egyptian patients with neck pain.

BACKGROUND:

Neck pain is a highly prevalent musculoskeletal disorders in adults affecting from 45.5% to 48%. It may cause disability that interferes with the quality of life. It is usually treated conservatively. To evaluate treatment effectiveness, patients need close monitoring and follow-up.

Different assessment tools are recommended including patient reported outcome measures. One of the newly introduced outcome measure is The Neck Core Outcome Measure Index (COMI). It is characterized by being brief, simple, self-reported and easy to answer questionnaire. The SPINE TANGO, which is the spine organization In Europe, has recommended its use for all patients with spine disorders.

This questionnaire has been translated into different languages such as German, Polish and Italian but it has never been translated and validated in the Arabic language.

HYPOTHESES

1. The Arabic version of neck-COMI will be a valid tool for the assessment of neck pain in Egyptian patients.
2. The Arabic version of neck-COMI will be a reliable tool for the assessment of neck pain in Egyptian patients.

RESEARCH QUESTION:

Will the Arabic version of neck-COMI be a valid and reliable tool to assess neck pain in the Egyptian patients?

DETAILED DESCRIPTION:
This study is translating and cross culturally adapting the COMI outcome measure for patients with neck pain in Egypt. This study will be conducted at the outpatient clinic of Cairo University hospitals in Egypt.

Translation:

The cross-cultural adaptation process for the COMI will be done as described by Beaton and colleagues (2000). This will include the following phases:

1. Initial translation that includes forward translation to translate the questionnaire from the English language to Arabic by two independent bilingual translators one of them is familiar with the concepts of the COMI and the other translator doesn't have medical background.
2. Synthesis of the translations by comparing the two Arabic translations and combine them into one version.
3. Back translation to translate the Arabic version to the English language again. This should be done by two independent translators both of them shouldn't have medical background, yet not familiar with the use of COMI then comparing between two backwards translations to determine any differences between them and the original one.
4. Expert committee that consists of both translators, one of the back-translators, one bilingual clinician and one native English clinical research scientist to compare between versions of the COMI and consolidate the final version. The role of the expert committee to detect and correct any conceptual errors or inconsistencies, grammatical or other errors.
5. Test of the pre-final version of the instrument in a small sample to assess its content and face validity according to patients' feedback and collect comments about wording and clarity of the translated version via semi-structured interview. This will be done in a sample of 20 patients who fulfill the study inclusion and exclusion criteria. Patients will be asked to complete the final Arabic version of COMI and will be asked to comment on any linguistic ambiguity. Finally, researcher will discuss received comments and a consensus will be done to adapt any necessary changes.

(2) Validation and reliability testing:

One hundred male and female adults will be recruited from physiotherapy and Orthopedic outpatient clinics.This sample size has been recommended as an appropriate size for reliability and validity analyses.

Validation testing:

COMI will be tested by comparing it with Visual Analogue scale (VAS), EuroQol-visual analogue scale (EQ-VAS), EuroQo-5D (EQ-5D), Neck disability index (NDI).

Reliability testing:

Each patient will be asked to complete the questionnaire booklet in two-separate sessions within 14 days.

ELIGIBILITY:
Inclusion Criteria:

1. Egyptian adult patients who are native Arabic speakers.
2. Age ranges from 20 and 60 years.
3. Referred with the diagnosis of chronic mechanical neck pain with and without arm pain.
4. Pain duration is greater than 3 months.

Exclusion Criteria:

1. Systemic diseases e.g. rheumatic diseases
2. Specific etiology of neck pain like spinal stenosis or fracture.
3. Previous surgery or trauma to the spine
4. Upper quadrant dysfunction, rather than radiculopathy.
5. Inability to read (illiterate)

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients will be selected from orthopedic and Physical therapy outpatient clinics
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2022-03-15 (Estimated)

PRIMARY OUTCOMES:
Concurrent validity | 1 day
  It will be established by correlating the COMI subsections to the relevant sections in the questionnaire booklet (that consists of the NDI, VAS, EQ-VAS, EQ-D5)

SECONDARY OUTCOMES:
Test-retest reliability | 5-14 days
  This will be examined by comparing the results between the Arabic COMI questionnaires filled in the two testing sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Aliaa Regan Youssef, PhD, Principal Investigator — Cairo University
Locations (1):
- Cairo university Outpatient clinics, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Andresen EM. Criteria for assessing the tools of disability outcomes research. Arch Phys Med Rehabil. 2000 Dec;81(12 Suppl 2):S15-20. doi: 10.1053/apmr.2000.20619. PMID 11128900
- [Background] Ariens GA, van Mechelen W, Bongers PM, Bouter LM, van der Wal G. Psychosocial risk factors for neck pain: a systematic review. Am J Ind Med. 2001 Feb;39(2):180-93. doi: 10.1002/1097-0274(200102)39:23.0.co;2-#. PMID 11170160
- [Background] Beaton DE, Bombardier C, Guillemin F, Ferraz MB. Guidelines for the process of cross-cultural adaptation of self-report measures. Spine (Phila Pa 1976). 2000 Dec 15;25(24):3186-91. doi: 10.1097/00007632-200012150-00014. No abstract available. PMID 11124735
- [Background] Blanpied PR, Gross AR, Elliott JM, Devaney LL, Clewley D, Walton DM, Sparks C, Robertson EK. Neck Pain: Revision 2017. J Orthop Sports Phys Ther. 2017 Jul;47(7):A1-A83. doi: 10.2519/jospt.2017.0302. PMID 28666405
- [Background] Bongers PM, Ijmker S, van den Heuvel S, Blatter BM. Epidemiology of work related neck and upper limb problems: psychosocial and personal risk factors (part I) and effective interventions from a bio behavioural perspective (part II). J Occup Rehabil. 2006 Sep;16(3):279-302. doi: 10.1007/s10926-006-9044-1. PMID 16850279
- [Background] Boonstra AM, Schiphorst Preuper HR, Reneman MF, Posthumus JB, Stewart RE. Reliability and validity of the visual analogue scale for disability in patients with chronic musculoskeletal pain. Int J Rehabil Res. 2008 Jun;31(2):165-9. doi: 10.1097/MRR.0b013e3282fc0f93. PMID 18467932
- [Background] Borghouts JAJ, Koes BW, Bouter LM. The clinical course and prognostic factors of non-specific neck pain: a systematic review. Pain. 1998 Jul;77(1):1-13. doi: 10.1016/S0304-3959(98)00058-X. PMID 9755013
- [Background] Cagnie B, Danneels L, Van Tiggelen D, De Loose V, Cambier D. Individual and work related risk factors for neck pain among office workers: a cross sectional study. Eur Spine J. 2007 May;16(5):679-86. doi: 10.1007/s00586-006-0269-7. Epub 2006 Dec 8. PMID 17160393
- [Background] Deyo RA, Battie M, Beurskens AJ, Bombardier C, Croft P, Koes B, Malmivaara A, Roland M, Von Korff M, Waddell G. Outcome measures for low back pain research. A proposal for standardized use. Spine (Phila Pa 1976). 1998 Sep 15;23(18):2003-13. doi: 10.1097/00007632-199809150-00018. PMID 9779535
- [Background] Drost, E. A. (2011). Validity and Reliability in Social Science Research. Education Research and Perspectives, 38(1), 105-123
- [Background] Dworkin RH, Turk DC, Farrar JT, Haythornthwaite JA, Jensen MP, Katz NP, Kerns RD, Stucki G, Allen RR, Bellamy N, Carr DB, Chandler J, Cowan P, Dionne R, Galer BS, Hertz S, Jadad AR, Kramer LD, Manning DC, Martin S, McCormick CG, McDermott MP, McGrath P, Quessy S, Rappaport BA, Robbins W, Robinson JP, Rothman M, Royal MA, Simon L, Stauffer JW, Stein W, Tollett J, Wernicke J, Witter J; IMMPACT. Core outcome measures for chronic pain clinical trials: IMMPACT recommendations. Pain. 2005 Jan;113(1-2):9-19. doi: 10.1016/j.pain.2004.09.012. No abstract available. PMID 15621359
- [Background] Eldridge S, Ashby D, Bennett C, Wakelin M, Feder G. Internal and external validity of cluster randomised trials: systematic review of recent trials. BMJ. 2008 Apr 19;336(7649):876-80. doi: 10.1136/bmj.39517.495764.25. Epub 2008 Mar 25. PMID 18364360
- [Background] Fankhauser CD, Mutter U, Aghayev E, Mannion AF. Validity and responsiveness of the Core Outcome Measures Index (COMI) for the neck. Eur Spine J. 2012 Jan;21(1):101-14. doi: 10.1007/s00586-011-1921-4. Epub 2011 Aug 20. PMID 21858567
- [Background] Feise RJ, Michael Menke J. Functional rating index: a new valid and reliable instrument to measure the magnitude of clinical change in spinal conditions. Spine (Phila Pa 1976). 2001 Jan 1;26(1):78-86; discussion 87. doi: 10.1097/00007632-200101010-00015. PMID 11148650
- [Background] Fejer R, Kyvik KO, Hartvigsen J. The prevalence of neck pain in the world population: a systematic critical review of the literature. Eur Spine J. 2006 Jun;15(6):834-48. doi: 10.1007/s00586-004-0864-4. Epub 2005 Jul 6. PMID 15999284
- [Background] Feng Y, Parkin D, Devlin NJ. Assessing the performance of the EQ-VAS in the NHS PROMs programme. Qual Life Res. 2014 Apr;23(3):977-89. doi: 10.1007/s11136-013-0537-z. Epub 2013 Oct 1. PMID 24081873
- [Background] Ferguson L. External validity, generalizability, and knowledge utilization. J Nurs Scholarsh. 2004;36(1):16-22. doi: 10.1111/j.1547-5069.2004.04006.x. PMID 15098414
- [Background] Guzman J, Hurwitz EL, Carroll LJ, Haldeman S, Cote P, Carragee EJ, Peloso PM, van der Velde G, Holm LW, Hogg-Johnson S, Nordin M, Cassidy JD. A new conceptual model of neck pain: linking onset, course, and care: the Bone and Joint Decade 2000-2010 Task Force on Neck Pain and Its Associated Disorders. J Manipulative Physiol Ther. 2009 Feb;32(2 Suppl):S17-28. doi: 10.1016/j.jmpt.2008.11.007. PMID 19251062
- [Background] Howard, H. (1996). The Quebec Task Force on Whiplash-Associated Disorders. Musculoskeletal Pain, 4(4), 95-104
- [Background] Hudswell, S., Von Mengersen, M., & Lucas, N. (2005). The cranio-cervical flexion test using pressure biofeedback : A useful measure of cervical dysfunction in the clinical setting ? International Journal of Osteopathic Medicine, 8(3), 98-105
- [Background] Jull, G. A. (2000). Deep Cervical Flexor Muscle Dysfunction in Whiplash. Musculoskeletal Pain, 8(1-2), 143-154
- [Background] Kaplan RM, Bush JW, Berry CC. Health status: types of validity and the index of well-being. Health Serv Res. 1976 Winter;11(4):478-507. PMID 1030700
- [Background] Kimberlin CL, Winterstein AG. Validity and reliability of measurement instruments used in research. Am J Health Syst Pharm. 2008 Dec 1;65(23):2276-84. doi: 10.2146/ajhp070364. PMID 19020196
- [Background] Klimek L, Bergmann KC, Biedermann T, Bousquet J, Hellings P, Jung K, Merk H, Olze H, Schlenter W, Stock P, Ring J, Wagenmann M, Wehrmann W, Mosges R, Pfaar O. Visual analogue scales (VAS): Measuring instruments for the documentation of symptoms and therapy monitoring in cases of allergic rhinitis in everyday health care: Position Paper of the German Society of Allergology (AeDA) and the German Society of Allergy and Clinical Immunology (DGAKI), ENT Section, in collaboration with the working group on Clinical Immunology, Allergology and Environmental Medicine of the German Society of Otorhinolaryngology, Head and Neck Surgery (DGHNOKHC). Allergo J Int. 2017;26(1):16-24. doi: 10.1007/s40629-016-0006-7. Epub 2017 Jan 19. PMID 28217433
- [Background] McHorney CA, Tarlov AR. Individual-patient monitoring in clinical practice: are available health status surveys adequate? Qual Life Res. 1995 Aug;4(4):293-307. doi: 10.1007/BF01593882. PMID 7550178
- [Background] McLean SM, May S, Klaber-Moffett J, Sharp DM, Gardiner E. Risk factors for the onset of non-specific neck pain: a systematic review. J Epidemiol Community Health. 2010 Jul;64(7):565-72. doi: 10.1136/jech.2009.090720. Epub 2010 May 12. PMID 20466711
- [Background] Miekisiak G, Banach M, Kiwic G, Kubaszewski L, Kaczmarczyk J, Sulewski A, Kloc W, Libionka W, Latka D, Kollataj M, Zaluski R. Reliability and validity of the Polish version of the Core Outcome Measures Index for the neck. Eur Spine J. 2014 Apr;23(4):898-903. doi: 10.1007/s00586-013-3129-2. Epub 2013 Dec 23. PMID 24363040
- [Background] Misailidou V, Malliou P, Beneka A, Karagiannidis A, Godolias G. Assessment of patients with neck pain: a review of definitions, selection criteria, and measurement tools. J Chiropr Med. 2010 Jun;9(2):49-59. doi: 10.1016/j.jcm.2010.03.002. PMID 21629550
- [Background] Misterska E, Jankowski R, Glowacki M. Cross-cultural adaptation of the Neck Disability Index and Copenhagen Neck Functional Disability Scale for patients with neck pain due to degenerative and discopathic disorders. Psychometric properties of the Polish versions. BMC Musculoskelet Disord. 2011 Apr 29;12:84. doi: 10.1186/1471-2474-12-84. PMID 21529360
- [Background] Monticone M, Ferrante S, Maggioni S, Grenat G, Checchia GA, Testa M, Teli MG, Mannion AF. Reliability, validity and responsiveness of the cross-culturally adapted Italian version of the core outcome measures index (COMI) for the neck. Eur Spine J. 2014 Apr;23(4):863-72. doi: 10.1007/s00586-013-3092-y. Epub 2013 Nov 23. PMID 24272267
- [Background] White P, Lewith G, Prescott P. The core outcomes for neck pain: validation of a new outcome measure. Spine (Phila Pa 1976). 2004 Sep 1;29(17):1923-30. doi: 10.1097/01.brs.0000137066.50291.da. PMID 15534418
- [Background] Rebbeck TJ, Refshauge KM, Maher CG, Stewart M. Evaluation of the core outcome measure in whiplash. Spine (Phila Pa 1976). 2007 Mar 15;32(6):696-702. doi: 10.1097/01.brs.0000257595.75367.52. PMID 17413477
- [Background] Sach TH, Barton GR, Doherty M, Muir KR, Jenkinson C, Avery AJ. The relationship between body mass index and health-related quality of life: comparing the EQ-5D, EuroQol VAS and SF-6D. Int J Obes (Lond). 2007 Jan;31(1):189-96. doi: 10.1038/sj.ijo.0803365. Epub 2006 May 9. PMID 16682976
- [Background] Schellingerhout JM, Verhagen AP, Heymans MW, Koes BW, de Vet HC, Terwee CB. Measurement properties of disease-specific questionnaires in patients with neck pain: a systematic review. Qual Life Res. 2012 May;21(4):659-70. doi: 10.1007/s11136-011-9965-9. Epub 2011 Jul 7. PMID 21735306
- [Background] Shaheen AA, Omar MT, Vernon H. Cross-cultural adaptation, reliability, and validity of the Arabic version of neck disability index in patients with neck pain. Spine (Phila Pa 1976). 2013 May 1;38(10):E609-15. doi: 10.1097/BRS.0b013e31828b2d09. PMID 23429690
- [Background] Stahl MK, El-Metwally AA, Mikkelsson MK, Salminen JJ, Pulkkinen LR, Rose RJ, Kaprio JA. Genetic and environmental influences on non-specific neck pain in early adolescence: a classical twin study. Eur J Pain. 2013 Jul;17(6):791-8. doi: 10.1002/j.1532-2149.2012.00247.x. Epub 2012 Nov 9. PMID 23139100
- [Background] Tawfik soliman, D. M. (2012). validity and reliability testing of translated arabic version of neck disability index
- [Background] Tsakitzidis, G., Remmen, R., Dankaerts, W., & Van Royen, P. (2013). Non- Specific Neck Pain and Evidence-Based Practice. European Scientific Journal (ESJ), 9(3), 1-19
- [Background] Turk DC, Dworkin RH, Revicki D, Harding G, Burke LB, Cella D, Cleeland CS, Cowan P, Farrar JT, Hertz S, Max MB, Rappaport BA. Identifying important outcome domains for chronic pain clinical trials: an IMMPACT survey of people with pain. Pain. 2008 Jul 15;137(2):276-285. doi: 10.1016/j.pain.2007.09.002. Epub 2007 Oct 15. PMID 17937976
- [Background] Vernon H. The Neck Disability Index: state-of-the-art, 1991-2008. J Manipulative Physiol Ther. 2008 Sep;31(7):491-502. doi: 10.1016/j.jmpt.2008.08.006. PMID 18803999
- [Background] Wainner RS, Fritz JM, Irrgang JJ, Boninger ML, Delitto A, Allison S. Reliability and diagnostic accuracy of the clinical examination and patient self-report measures for cervical radiculopathy. Spine (Phila Pa 1976). 2003 Jan 1;28(1):52-62. doi: 10.1097/00007632-200301010-00014. PMID 12544957
- [Background] Ware JE Jr. SF-36 health survey update. Spine (Phila Pa 1976). 2000 Dec 15;25(24):3130-9. doi: 10.1097/00007632-200012150-00008. No abstract available. PMID 11124729
- [Background] Whynes DK; TOMBOLA Group. Correspondence between EQ-5D health state classifications and EQ VAS scores. Health Qual Life Outcomes. 2008 Nov 7;6:94. doi: 10.1186/1477-7525-6-94. PMID 18992139